CLINICAL TRIAL: NCT04601090
Title: Survival Rates and Long-term Outcomes for Patients With COVID-19 Admitted to Norwegian ICUs
Brief Title: Survival Rates and Longterm Outcomes After COVID-19
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Kristin Hofsø, PhD, Oslo University Hospital
Other Study IDs: 135310
Record Dates: First submitted 2020-10-15; First posted 2020-10-23 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Acute Respiratory Failure; Acute Respiratory Distress Syndrome; Post Intensive Care Unit Syndrome; Survivorship
Keywords: ICU treatment
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ICU treatment — This is an observational study, so all patients will undergo a variation of ICU treatment, and we will record that information (e.g., time on ventilator, time in ICU, SAPS score at admission)

SUMMARY:
The study 'Survival rates and long-term outcomes for patients with COVID-19 admitted to Norwegian ICUs' is a national observational study, including patients admitted to a Norwegian ICU between March 2020 and March 2021. The study will describe survival rates, clinical characteristics and health challenges experienced by survivors the first year after ICU admission caused by COVID-19 disease.

DETAILED DESCRIPTION:
The study 'Survival rates and long-term outcomes for patients with COVID-19 admitted to Norwegian ICUS' has two different aims. The first aim is to synthesis data from a National register (Norwegian Intensive care register-NIR) on all COVID-19 patients in Norway admitted to an ICU. These results are of great public interest for many reasons. First of all, it will give us information on the severity of this novel virus, but also how the health care system has coped in treating the severe cases that was admitted to an ICU. The results will potentially be compared to other patient populations with viral pneumonia, but most interestingly to survival rates from other countries. In addition, the data will give us a description on how the distribution of severe cases of COVID-19 have been within Norway (e.g., gender, age, health regions etc.) The second aim of this study is to measure and describe health related challenges COVID-19 patients may experience during their first year from ICU admission. The health-related domains that will be investigated will capture both mental, physical and cognitive health. Knowledge from other patient population admitted to an ICU with acute respiratory failure, indicates that these are the main domains that negatively affect the activity of daily living. Physical, mental and cognitive health challenges will be investigated for the Norwegian COVID -19 population admitted to ICU, and will give important insight to the impact COVID-19 can have on survivors of severe cases, as well as the need for rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered in Norwegian Intensive Care Register, that are ≥ 18 years with confirmed cases of COVID-19.

Exclusion Criteria:

* Exclusion criteria only for follow-up study: Do not understand Norwegian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that have been admitted to a Norwegian ICU with confirmed COVID-19, and not reserved them against the national register, will be contacted for inclusion to the study.
Sampling Method: Non-Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
ICU Survival rate | up to 30 days
  Time to survival
Change in Functional Status | 6 and 12 months after ICU admission
  Measured by self-reporting using Lawton Instrumental activity of daily living. Higher score indicates better function, and ranges from 0-8.

SECONDARY OUTCOMES:
Change in Anxiety and Depression | Measured 6 and 12 months after ICU admission
  Measured by self-report using Hospital Anxiety and Depression Scale (HADS). Higher score indicates higher lever of anxiety and depression, scored on separate sub scales (0-21 for each).
Changes in Cognitive Status | Measured at 6 and 12 months after ICU admission
  Measured by telephone interview using the Mini Montreal Cognitive Assessment, score ranges from 0-15. Higher score indicates better cognitive function.
Change in Quality of Life 6 and 12 months after ICU admission | Measured 6 and 12 months after ICU admission
  Measured by self report using (Euroqual 5 dimensions) EQ-5D. Higher score indicates worse health (range 5-15).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Hofsø, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laake JH, Hagen M, Aavitsland P, Buanes EA, Fjone KS, Kvale R, Olsen BF, Hofso K. COVID-19 in Norwegian ICUs 2020-2023: Patient characteristics, management, and outcomes-A nationwide prospective observational study. Acta Anaesthesiol Scand. 2025 Apr;69(4):e70027. doi: 10.1111/aas.70027. PMID 40114460